CLINICAL TRIAL: NCT01723163
Title: Abstinence Reinforcement Therapy (ART) for Rural Veteran Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 12-365
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Veteran; Smoking Cessation
Keywords: veteran; smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Methods; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Abstinence Reinforcement Therapy (ART)
  Interventions: Behavioral: Abstinence Reinforcement Therapy (ART)
- Control (Other): Telephone Counseling
  Interventions: Behavioral: Telephone Counseling and NRT

INTERVENTIONS:
Behavioral: Abstinence Reinforcement Therapy (ART) — Veterans randomized to the intervention will receive cognitive-behavioral telephone counseling (TC), a tele-medicine clinic for access to nicotine replacement (NRT), and mobile contingency management (mCM)
  Other Names: Intervention
  Arms: Intervention
Behavioral: Telephone Counseling and NRT — Veterans randomized to the control group will receive cognitive-behavioral telephone counseling (TC) and a tele-medicine clinic for access to nicotine replacement (NRT)
  Other Names: Control
  Arms: Control

SUMMARY:
The primary goal of the current study is to evaluate the effectiveness of a combined tele-health and contingency management (CM) intervention that investigators are calling Abstinence Reinforcement Therapy (ART). Proposed is a comparative effectiveness trial with a two-group design in which 310 Veteran smokers will be randomized to either:

ABSTINENCE REINFORCEMENT THERAPY (ART) a proactive tele-health intervention that combines guideline based cognitive-behavioral telephone counseling (TC), a tele-medicine clinic for access to nicotine replacement (NRT), and intensive behavioral therapy through mobile contingency management.

TELE-HEALTH FOR SMOKING CESSATION a proactive tele-health intervention that will provide controls for therapist, medication, time and attention effects. The tele-health intervention provides the same guideline based cognitive-behavioral smoking cessation telephone counseling (TC), and tele-medicine clinic for access to NRT as in the ART intervention.

DETAILED DESCRIPTION:
The addition of contingency management (CM) to existing evidenced-based tele-health smoking cessation interventions is expected to be a cost-effective way to increase the reach of intensive smoking cessation treatment. CM is an intensive behavioral therapy that provides positive reinforcers (e.g., money, vouchers) to individuals misusing substances contingent upon objective evidence of abstinence from drug use. Implementation of CM has been limited because of the need to verify abstinence multiple times daily with a clinic based carbon monoxide (CO) monitor. As a result, CM approaches have largely been relegated to inpatient and day treatment programs. The application of emerging smart-phone technology, however, can overcome this barrier. Investigators have developed a smart-phone application which allows a participant to video themselves several times daily while using a small CO monitor and to transmit the data to a secure server. This innovation has made the use of CM for outpatient smoking cessation portable and feasible, i.e., mobile CM (mCM). Thus, the primary goal of the current study is to evaluate the effectiveness of a combined tele-health and CM intervention that investigators are calling Abstinence Reinforcement Therapy (ART). Proposed is a comparative effectiveness trial with a two-group design in which 310 Veteran smokers will be randomized to either:

ABSTINENCE REINFORCEMENT THERAPY (ART) a proactive tele-health intervention that combines guideline based cognitive-behavioral telephone counseling (TC), a tele-medicine clinic for access to nicotine replacement (NRT), and intensive behavioral therapy through mobile contingency management.

TELE-HEALTH FOR SMOKING CESSATION a proactive tele-health intervention that will provide controls for therapist, medication, time and attention effects. The tele-health intervention provides the same guideline based cognitive-behavioral smoking cessation telephone counseling (TC), and tele-medicine clinic for access to NRT as in the ART intervention.

Both of the proposed interventions are designed in accordance with national smoking cessation guidelines. Tele-health smoking cessation interventions are typically less intensive than clinic based specialty care, but increase reach of services through bypassing barriers to participation such as geographical distance from VA care. The addition of mCM to an evidence-based tele-health smoking intervention will significantly increase the intensity of the intervention and is predicted to increase efficacy. If cessation programs are to have significant impact (Impact = Reach X Efficacy) on changing health behavior at the population level, investigators must identify new and innovative strategies to increase treatment intensity, access, and participation.

The primary aim is to evaluate the impact of ART on rates of abstinence from cigarettes at 3-month, 6-month, and 12-month post-randomization follow-ups.

Hypothesis 1: Abstinence rates will be significantly higher among Veterans randomized to the ART-based intervention than those randomized to the Tele-health alone intervention (primary end-point; self-reported and bio-verified prolonged abstinence at the 6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Durham VA for ongoing care.
* Current smokers planning to quit smoking in the next 30 days.

Exclusion Criteria:

* Active diagnosis of psychosis documented in the medical record.
* Does not have access to a telephone.
* Severely impaired hearing or speech (Veterans must be able to respond to phone calls).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Calhoun, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wilson SM, Hair LP, Hertzberg JS, Kirby AC, Olsen MK, Lindquist JH, Maciejewski ML, Beckham JC, Calhoun PS. Abstinence Reinforcement Therapy (ART) for rural veterans: Methodology for an mHealth smoking cessation intervention. Contemp Clin Trials. 2016 Sep;50:157-65. doi: 10.1016/j.cct.2016.08.008. Epub 2016 Aug 10. PMID 27521811
- [Result] Dennis PA, Kimbrel NA, Dedert EA, Beckham JC, Dennis MF, Calhoun PS. Supplemental nicotine preloading for smoking cessation in posttraumatic stress disorder: Results from a randomized controlled trial. Addict Behav. 2016 Aug;59:24-9. doi: 10.1016/j.addbeh.2016.03.004. Epub 2016 Mar 11. PMID 27046670
- [Result] Green KT, Wilson SM, Dennis PA, Runnals JJ, Williams RA, Bastian LA, Beckham JC, Dedert EA, Kudler HS, Straits-Troster K, Gierisch JM, Calhoun PS. Cigarette Smoking and Musculoskeletal Pain Severity Among Male and Female Afghanistan/Iraq Era Veterans. Pain Med. 2017 Sep 1;18(9):1795-1804. doi: 10.1093/pm/pnw339. PMID 28340108
- [Result] Calhoun PS, Wilson SM, Hertzberg JS, Kirby AC, McDonald SD, Dennis PA, Bastian LA, Dedert EA; VA Mid-Atlantic MIRECC Workgroup; Beckham JC. Validation of Veterans Affairs Electronic Medical Record Smoking Data Among Iraq- and Afghanistan-Era Veterans. J Gen Intern Med. 2017 Nov;32(11):1228-1234. doi: 10.1007/s11606-017-4144-5. Epub 2017 Aug 14. PMID 28808856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who did not complete a follow-up were not prohibited from participating in the remaining study follow-up periods.
Period: Baseline
Arm/Group | Intervention | Control
Started | 156 | 154
Completed | 156 | 154
Not Completed | 0 | 0
Period: Treatment Phase
Arm/Group | Intervention | Control
Started | 156 | 154
Completed | 137 | 147
Not Completed | 19 | 7
Not completed — Withdrawal by Subject | 14 | 6
Not completed — Withdrawal by PI | 5 | 1
Period: 3-Month Follow-up
Arm/Group | Intervention | Control
Started | 137 | 147
Completed | 124 | 128
Not Completed | 13 | 19
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unable to Contact | 12 | 19
Period: 6-Month Follow-up
Arm/Group | Intervention | Control
Started | 136 | 147
Completed | 118 | 132
Not Completed | 18 | 15
Not completed — Death | 1 | 0
Not completed — Unable to Contact | 17 | 15
Period: 12-Month Follow-up
Arm/Group | Intervention | Control
Started | 135 | 147
Completed | 111 | 119
Not Completed | 24 | 28
Not completed — Death | 1 | 0
Not completed — Unable to Contact | 23 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 156 | 154 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11) | 56 (11) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 139 | 137 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 153 | 152 | 305
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 90 | 175
  White | 61 | 56 | 117
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  More than High School | 101 | 103 | 204
  High School or less | 55 | 51 | 106
Distance to nearest VA hospital or clinic (miles) [Count of Participants; unit: Participants] — Distance from the participant's home to the nearest VA hospital or VA clinic (in miles).
  Participants
    0-20 Miles | 56 | 53 | 109
    21-40 Miles | 49 | 66 | 115
    41-60 Miles | 35 | 21 | 56
    61-80 Miles | 9 | 6 | 15
    81-100 Miles | 5 | 5 | 10
    101 Miles or more | 2 | 3 | 5
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Scores can range from 0-10; higher scores reflect a higher level of nicotine dependence.
  units on a scale | 4 (2) | 4 (2) | 4 (2)
Self efficacy scale for quitting smoking in next 6 months [Mean (Standard Deviation); unit: units on a scale] — 1=not at all to 7=very confident
  units on a scale | 6 (1) | 6 (1) | 6 (1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abstinence or Non-Abstinence at 6-month Follow-up
Description: Non-abstinence is defined as smoking for 7 consecutive days or at least once a week for 2 consecutive weeks. Non-abstinence was evaluated for the 90 days previous to the 6 month follow-up.
Time Frame: 6-month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 156 | 154
Participants
  Abstinent | 38 | 40
  Non-Abstinent | 77 | 83
  Missing | 41 | 31

ADVERSE EVENTS:
Time Frame: up to 12 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/156 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/154
Other Adverse Events (participants affected / at risk) | 0/156 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No